CLINICAL TRIAL: NCT05538962
Title: Longitudinal Monitoring of Inflammation in Cirrhosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BAJAJ0028
Record Dates: First submitted 2022-09-07; First posted 2022-09-14 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Cirrhosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Intervention Model Description: All subjects will receive the sensor but they are 3 different populations, which is why there are 3 different arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy controls (Experimental): Healthy controls will receive the sensors
  Interventions: Diagnostic Test: Sensor skin
- Outpatients with cirrhosis (Experimental): Outpatients with cirrhosis will receive the sensors
  Interventions: Diagnostic Test: Sensor skin
- Inpatients with cirrhosis (Experimental): Inpatients with cirrhosis will receive the sensors
  Interventions: Diagnostic Test: Sensor skin

INTERVENTIONS:
Diagnostic Test: Sensor skin — Skin sensor to detect inflammatory molecules in sweat

SUMMARY:
Longitudinal monitoring of inflammation using skin devices may help predict outcomes compared to traditional blood draws

ELIGIBILITY:
Healthy Volunteers

Inclusion Criteria:

1. Age >18 years
2. Able to give consent

Exclusion Criteria:

1. Unable/unwilling to consent
2. Chronic diseases
3. Unable to come in daily or be available daily for 3 days.

Outpatients with Cirrhosis:

Inclusion criteria:

1. Age >18 years
2. Able to give consent
3. Cirrhosis defined by any one of the following

   1. Cirrhosis on liver biopsy or transient wave elastography
   2. Nodular liver on imaging
   3. Endoscopic or radiological evidence of varices in a patient with chronic liver disease
   4. Platelet count <150,000/mm3 and AST/ALT ratio >1 in a patient with chronic liver disease
   5. Patients with frank decompensation (ascites, HE, variceal bleeding, hepato-pulmonary syndrome)

Exclusion criteria:

1. Unable/unwilling to consent
2. Unclear diagnosis of cirrhosis
3. Unable to come in daily or be available daily for 3 days.
4. Inflammatory bowel disease or other diseases that require immunosuppressive therapy use

Inpatients with Cirrhosis:

Inclusion criteria:

1. Age >18 years
2. Able to give consent
3. Cirrhosis defined by any one of the following

   1. Cirrhosis on liver biopsy or transient wave elastography
   2. Nodular liver on imaging
   3. Endoscopic or radiological evidence of varices in a patient with chronic liver disease
   4. Platelet count <150,000/mm3 and AST/ALT ratio >1 in a patient with chronic liver disease
   5. Patients with frank decompensation (ascites, HE, variceal bleeding, hepato-pulmonary syndrome)

Exclusion criteria:

1. Unable/unwilling to consent
2. Unclear diagnosis of cirrhosis
3. Unable to be seen daily or able to come in daily for 3 days (if discharged in between)
4. Inflammatory bowel disease or other diseases that require immunosuppressive therapy use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 days
  We will study whether subjects have any issues or adverse events related to the sensor

SECONDARY OUTCOMES:
Ability to detect inflammatory markers (TNF, IL-1b, IL-6 and CRP) using skin sensor compared to blood values | 3 days
  Comparison of skin sensor data to blood inflammatory markers as above using daily blood draw and sensor values. Blood markers and sensor markers will be correlated for each day.
Linkage of skin inflammatory markers (TNF, IL-6, IL-1b and CRP) with quality of life | 3 days
  Correlation of inflammatory markers using the skin sensor data to quality of life using Sickness Impact Profile and PROMIS questionnaires.
Linkage of inflammatory markers (TNF, IL-6, IL-1b and CRP) with cognitive testing | 3 days
  Correlation of inflammatory markers using the skin sensor data to cognitive performance on PHES and EncephalApp Stroop
Linkage of inflammatory markers with MELD score | 3 days
  Correlation of inflammatory markers using the skin sensor data to MELD score

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan Bajaj, MD, Principal Investigator — Hunter Holmes McGuire VAMC
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No